CLINICAL TRIAL: NCT02510417
Title: Administration of Most Closely HLA-matched Multivirus-specific Cytotoxic T-Lymphocytes for the Treatment of EBV, CMV, Adenovirus Infections Post Allogeneic Stem Cell Transplant
Brief Title: Allogeneic Virus-specific T Cell Lines (VSTs)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director- Program for Cell Enhancement and Technologies for Immunotherapy (CETI), Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHAPS
Record Dates: First submitted 2015-07-13; First posted 2015-07-29 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Viral Infections After HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- VSTs against three viruses (Experimental): Patients will receive 2 x 107 partially HLA-matched VSTs/m2 as a single infusion. In the rare case where insufficient banked cell product is available, a lower number of cells may be infused after discussion with the principal investigator, patient and/or guardian and the treatment team. If participants have a partial response (as defined by a 50% fall in viral load) they are eligible to receive up to 4 additional doses from day 28 after the initial infusion and at 2 weekly intervals thereafter.
  Interventions: Biological: VSTs

INTERVENTIONS:
Biological: VSTs — most closely HLA-matched multivirus-specific T cell lines obtained from a bank of allogeneic virus-specific T cell lines (VSTs) have antiviral activity against three viruses: EBV, CMV and adenovirus

SUMMARY:
The primary purpose of the study is to evaluate whether most closely HLA-matched multivirus-specific T cell lines obtained from a bank of allogeneic virus-specific T cell lines (VSTs) have antiviral activity against three viruses: EBV, CMV and adenovirus.

Reconstitution of anti-viral immunity by donor-derived VSTs has shown promise in preventing and treating infections associated with CMV, EBV and adenovirus post-transplant. However, the time taken to prepare patient-specific products and lack of virus-specific memory T cells in cord blood and seronegative donors, limits their value.

An alternative is to use banked partially HLA-matched allogeneic VSTs. A prior phase II study at our institution using trivirus-specific VSTs generated using monocytes and EBV-transformed B cells gene-modified with a clinical grade adenoviral vector expressing CMV-pp65 to activate and expand specific T cells showed the feasibility, safety and activity of this approach for the treatment of refractory CMV, EBV and Adenovirus infections. However, the production process was lengthy, requiring 8-12 weeks, with exposure to biohazards (B95.8 EBV viral strain and adenovector), while antigenic competition between different viral components precluded increasing the spectrum of specificity beyond these three viruses.

Investigator have overcome these limitations and in the current trial, they will evaluate whether rapidly generated, allogeneic most closely HLA-matched multivirus-specific VSTs, activated using overlapping peptide libraries spanning immunogenic antigens from CMV, adenovirus and EBV will be safe and produce anti-viral effects in allogeneic HSCT recipients infected with one of more of the targeted viruses that are persistent despite conventional anti-viral therapy. The study agent will be assessed for safety (stopping rules defined) and antiviral activity.

DETAILED DESCRIPTION:
Investigators evaluated the clinical utility of Multivirus VSTs in recipients of matched related, matched unrelated, or haploidentical donor transplants. To date, 10 clinical-grade multivirus-directed VSTs have been generated from donor PBMCs. These lines were polyclonal, comprising both CD4+ (57±5%) and CD8+ (35±5%) cells and retained expression of the memory markers CD45RO+CD62L+ (58±8%). Their specificity was dependent on the prior viral exposure of the cell donor; 7/8 tested lines had activity against Adv,8/8 against CMV, 6/8 against EBV. None of the lines reacted against recipient PHA blasts - indicating lack of alloreactive potential in these rapidly generated lines.

Investigators administered these multivirus-specific donor-derived VSTs to 3 allogeneic HSCT recipients in a dose escalation study all on DL1 (5x106/m2). There were no immediate infusion toxicities, and no de novo acute GvHD, demonstrating the in vivo safety of these mVST. Further, antiviral efficacy has been observed in 1 patient with refractory CMV. In addition, in a recently published paper from Baylor College of Medicien (Anapoulous et al, STM 2014) they have treated VSTs manufactured with a similar methodology, but targeting 5 viruses instead of 3 with specificity to BK virus and HHV6. In that study 10 patients were treated with 4 on DL1 (5x10e6/m2), 4 on DL2 (1x10e7/m2) and 2 on DL3 (2x10e7/m2) and again saw no immediate infusion toxicities, and no de novo acute GvHD, demonstrating the in vivo safety of these mVST. Three patients received the cells as viral prophylaxis (days 38-43 post-HSCT) and none developed viral infections at up to 3 months post-treatment. The other 7 patients received the cells as treatment for one or more active infections between days 59-139 post-HSCT. Based on viral load measurements by day 42 post-infusion, the VSTs were successful in controlling active infections with CMV (1 complete (CR) and 1 partial response (PR)), EBV (2 CRs, including a case of frank PTLD); Adv (1 CR); HHV6 (1 CR); and BK (3 CR, 1 PR, 1NR). Of note, 3 BK virus responders had tissue disease with severe hemorrhagic cystitis and all had marked improvement or disappearance of hematuria following infusion. One patient subsequently had an episode of transient but severe bladder pain in association with inflammation seen on cytoscopy coincident with a 6 log fall in urine BK viral load. Only non-responder was a patient with BK infection whose line lacked activity for this virus, likely reflecting the serostatus of the donor. In addition, 3 patients subsequently reactivated other viruses than those for which they were initially treated, but all cleared these infections by week 12, without the requirement for additional cell infusions (CMV: 1CR; EBV: 1CR; BK: 1CR; HHV6: 1CR). Finally, 1 patient received multivirus specific VSTs under a single patient protocol as an emergency treatment for widespread and bulky rituximab-resistant EBV-PTLD. Post VST treatment there was an immediate decline in the patient's EBV viral load with complete and sustained resolution of PTLD, coincident with an increase in circulating EBV-specific T cells. However, the profound anti-tumor activity mediated by the rapidly-expanding EBV-directed T cells also produced a transient systemic inflammatory response syndrome, which was controlled with steroids and anti-TNFR antibody, with no long term adverse effects.

Thus, infusion of donor-derived, multivirus specific VSTs generated with clinical grade pepmixes and infused either prophylactically or as treatment for one or more viral infections has been safe and is associated with the appearance of virus-reactive T cells in peripheral blood that have been able to control infection with above mentioned viruses.

ELIGIBILITY:
Inclusion Criteria:

1. Received prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow, single/double cord blood or PBSC
2. Cells administered as;

   1. Treatment of persistent or relapsed reactivation or infection
   2. Early treatment for single or multiple infections with EBV, CMV and/or adenovirus
3. Steroids less or equal to 0.5 mg/kg/day prednisone

5)Bilirubin <3x, AST <3x, Serum creatinine <2x upper limit of normal, Hgb >8.0, plts >20 6) Pulse oximetry of > 90% on room air 7) Available VSTs 8) Negative pregnancy test (if female of childbearing potential after reduced intensity conditioning) 9) Patient or parent/guardian capable of providing informed consent.

Exclusion Criteria:

1. Received ATG, Campath or other T cell immunosuppressive monoclonal antibodies in the last 28 days.
2. Patients with other uncontrolled infections
3. Received donor lymphocyte infusion in last 28 days
4. Evidence of GVHD > or equal to grade 2
5. Active and uncontrolled relapse of malignancy

Ages: 4 Weeks to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Assessments of patients with adverse events after VSTs infusion. | 45 days
  Safety of administration of VSTs is 45 days for GVHD. The safety endpoint will be defined as acute GvHD grades III-IV related to the T cell product within 45 days of the last VST dose and that are not due to the pre-existing infection or the original malignancy or pre-existing co-morbidities as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Assessments of viral load response to the CTL infusion | 12 months
  Increase in viral load of at least 50% from baseline or dissemination to other sites of disease.
Assessments of Antiviral Immunity | 12 months
  Patient serum and peripheral blood mononuclear cells will be monitored for virus-specific activity by phenotypic and functional studies including ELIspot with appropriate viral specific peptide mixtures and available HLA-restricted epitope peptides, intracellular cytokine staining, serum cytokine profiling and/or other assays as they become available for immune profiling purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bollard, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States